CLINICAL TRIAL: NCT02714569
Title: A Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Oral Ascending Dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of LY3202328
Brief Title: A Study to Evaluate LY3202328 in Overweight Healthy Participants and Dyslipidemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16417; I8Q-MC-GSEA (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-03-16; First posted 2016-03-21 (Estimated); Results first posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Dyslipidemias
MeSH Terms: conditions — Dyslipidemias | interventions — Atorvastatin; Simvastatin

STUDY DESIGN:
Intervention Model Description: Part A is a crossover. Part B is a parallel assignment.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part A: LY3202328 (LY) (Experimental): Single ascending doses of 1 milligram (mg), 3 mg, 10 mg, 30 mg, 100 mg, 300mg, 600 mg LY3202328 orally while fasting, or 30 mg LY3202328 orally while fed in 4 periods.
  Interventions: Drug: LY3202328
- Part A: Placebo (Placebo Comparator): A single ascending dose of placebo orally, in 1 period while fasting, and up to one period while fed.
  Interventions: Drug: Placebo
- Part B: LY3202328 (LY) (Experimental): A multiple ascending dose of 5 mg, 20 mg, 100 mg, and 300 mg LY3202328 at up to 4 dose levels, orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (atorvastatin or simvastatin) one week prior to treatment and on Day 29.
  Interventions: Drug: LY3202328; Drug: Atorvastatin; Drug: Simvastatin
- Part B: Placebo (Placebo Comparator): A multiple ascending dose of placebo at up to 4 dose levels, orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (atorvastatin or simvastatin) one week prior to treatment and on Day 29.
  Interventions: Drug: Placebo; Drug: Atorvastatin; Drug: Simvastatin

INTERVENTIONS:
Drug: LY3202328 — Administered orally
  Arms: Part A: LY3202328 (LY); Part B: LY3202328 (LY)
Drug: Placebo — Administered orally
  Arms: Part A: Placebo; Part B: Placebo
Drug: Atorvastatin — Administered orally
  Arms: Part B: LY3202328 (LY); Part B: Placebo
Drug: Simvastatin — Administered orally
  Arms: Part B: LY3202328 (LY); Part B: Placebo

SUMMARY:
The purpose of this two-part study is to evaluate the safety and tolerability of the study drug known as LY3202328 in healthy overweight participants in Part A, and those with dyslipidemia (abnormal blood fats) in Part B.

ELIGIBILITY:
Inclusion Criteria:

* Be healthy, as determined by medical history and physical examination
* Male participants must be between 18 and 70 years of age and must agree to use a reliable method of birth control during the study and 3 months following the last dose of the investigational product
* Female participants must be between 40 and 70 years old, and either postmenopausal or with a hysterectomy, and not pregnant and not lactating
* Be on a stable diet and exercise regimen for greater than (>) 3 months prior
* Have a body mass index (BMI) of 25.0 to 35.0 (Part A) or 27.0 to 40.0 (Part B) kilograms per meter squared
* Have fasting triglycerides (TG) between 150 and 499 milligrams per deciliter (mg/dL) (Part B only)
* Have a fasting low-density lipoprotein cholesterol (LDL-c) between 100 and 200 mg/dL (Part B only)
* Have estimated glomerular filtration rate greater than or equal to (≥) 60 milliliters per minute/1.73 meter squared with no proteinuria
* Be normotensive defined as supine systolic blood pressure (BP) less than or equal to (≤) 150 millimeters of mercury (mm Hg) and diastolic BP ≤ 100 mm Hg, without the use of any antihypertensive

Exclusion Criteria:

* Are taking a statin, any proprotein convertase subtilisin/kexin type 9 (PCSK9) medications, or have started taking other TG lowering agents (for example, niacin, fish oils)
* Are currently enrolled in a clinical trial involving an investigational product or off-label use of a drug or device, or are concurrently enrolled in any other type of medical research, or have participated in a clinical trial involving an investigational product or non-approved use of a drug within the last 30 days or within 5 half-lives
* Have an abnormal electrocardiogram or corrected QT or are on antihypertensive treatment
* Have any current or prior history of significant cardiovascular disease
* Show evidence of hepatitis C virus (HCV), Hepatitis B or other chronic liver disease
* Have an alcohol intake that exceeds 7 units per week with no more than 3 units per day, or are unwilling to stop alcohol consumption for the duration of the study (1 unit = 12 ounces or 360 mL of beer; 5 ounces or 150 mL of wine; 1.5 ounces or 45 mL of distilled spirits), or are a regular user of known drugs of abuse
* Have a history of untreated endocrine illness such as diabetes mellitus
* Have been on medications or supplements for weight loss within 3 months
* Have a history of active neuropsychiatric disease or on pharmacological therapy for such conditions (Part B, only)
* Show evidence of human immunodeficiency virus (HIV) infection
* Have been on medications that are known to inhibit cytochrome P450, family 3, subfamily A (CYP3A) or P-glycoprotein (P-gp), or regularly consume grapefruit
* Have donated blood of more than 500 mL within the last month
* Smoke >10 cigarettes per day or are unwilling to follow smoking rules

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03; Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- United States (4):
  - Clinical Pharmacology of Miami, Inc., Miami, Florida
  - PRA Health Sciences, Lenexa, Kansas
  - PRA Health Sciences, Marlton, New Jersey
  - PRA Health Sciences, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3202328 in Overweight Healthy Participants and in Participants With Dyslipidemia — https://www.lillytrialguide.com/en-US/studies/dyslipidemia/GSEA#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part A participants were divided into 2 cohorts. Within each cohort, participants were randomized to a treatment sequence (4 periods; up to 3 LY dose levels and at least one placebo). A 2-week washout occurred between each period. Part B participants were divided into 4 cohorts. Within each cohort, participants were randomized to LY or placebo.
Groups:
- Part A: Cohort 1(C1), Sequence 1: 1 milligram (mg) of LY3202328 (LY) was taken orally first intervention, then 10 mg of LY was taken orally second intervention, then placebo was taken orally third intervention, then 600 mg of LY was taken orally fourth intervention.
  C1, Sequence 1: (1 mg LY, 10 mg LY, Placebo, 600 mg LY)
- Part A: C1, Sequence 2: 1 mg of LY was taken orally first intervention, then placebo was taken orally second intervention, then 100 mg of LY was taken orally third intervention, then 600 mg of LY was taken orally fourth intervention.
  C1, Sequence 2: (1 mg LY, Placebo, 100 mg LY, 600 mg LY)
- Part A: C1, Sequence 3: Placebo was taken orally first intervention, then 10 mg LY was taken orally second intervention, then, 100 mg LY was taken orally third intervention, then placebo was taken orally fourth intervention.
  C1, Sequence 3: (Placebo, 10 mg LY, 100 mg LY, Placebo)
- Part A: Cohort 2 (C2), Sequence 1: 3 mg of LY was taken orally first intervention, then 30 mg of LY was taken orally second intervention, then placebo was taken orally third intervention, then 30 mg of LY fed was taken orally fourth intervention.
  C2, Sequence 1: (3 mg LY, 30 mg LY, Placebo, 30 mg LY Fed)
- Part A: C2, Sequence 2: 3 mg of LY was taken orally first intervention, then placebo was taken orally second intervention, then 300 mg of LY was taken orally third intervention, then placebo was taken orally fourth intervention.
  C2, Sequence 2: (3 mg LY, Placebo, 300 mg LY, Placebo)
- Part A: C2, Sequence 3: Placebo was taken orally first intervention, then 30 mg of LY was taken orally second intervention, then 300 mg of LY was taken orally third intervention, then 30 mg of LY fed was taken orally fourth intervention.
  C2, Sequence 3: (Placebo, 30 mg LY, 300 mg LY, 30 mg LY Fed)
- Part B: C3 (Simvastatin [SS]/Atorvastatin[AS] + 5 mg LY): 5 mg of LY was taken orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29.
- Part B: C4 (SS/AS + 20 mg LY): 20 mg of LY was taken orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29.
- Part B: C5 (SS/AS + 100 mg LY): 100 mg of LY was taken orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29.
- Part B: C6 (SS/AS + 300 mg LY): 300 mg of LY was taken orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29.
- Part B: C3-C6 (SS/AS + Placebo): Participants were randomly assigned to multiple ascending doses of placebo instead of LY at up to 4 dose levels, orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29.
Period: Part A First Intervention
Arm/Group | Part A: Cohort 1(C1), Sequence 1 | Part A: C1, Sequence 2 | Part A: C1, Sequence 3 | Part A: Cohort 2 (C2), Sequence 1 | Part A: C2, Sequence 2 | Part A: C2, Sequence 3 | Part B: C3 (Simvastatin [SS]/Atorvastatin[AS] + 5 mg LY) | Part B: C4 (SS/AS + 20 mg LY) | Part B: C5 (SS/AS + 100 mg LY) | Part B: C6 (SS/AS + 300 mg LY) | Part B: C3-C6 (SS/AS + Placebo)
Started | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Second Intervention
Arm/Group | Part A: Cohort 1(C1), Sequence 1 | Part A: C1, Sequence 2 | Part A: C1, Sequence 3 | Part A: Cohort 2 (C2), Sequence 1 | Part A: C2, Sequence 2 | Part A: C2, Sequence 3 | Part B: C3 (Simvastatin [SS]/Atorvastatin[AS] + 5 mg LY) | Part B: C4 (SS/AS + 20 mg LY) | Part B: C5 (SS/AS + 100 mg LY) | Part B: C6 (SS/AS + 300 mg LY) | Part B: C3-C6 (SS/AS + Placebo)
Started | 3 | 3 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 3 | 2 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 2 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Third Intervention
Arm/Group | Part A: Cohort 1(C1), Sequence 1 | Part A: C1, Sequence 2 | Part A: C1, Sequence 3 | Part A: Cohort 2 (C2), Sequence 1 | Part A: C2, Sequence 2 | Part A: C2, Sequence 3 | Part B: C3 (Simvastatin [SS]/Atorvastatin[AS] + 5 mg LY) | Part B: C4 (SS/AS + 20 mg LY) | Part B: C5 (SS/AS + 100 mg LY) | Part B: C6 (SS/AS + 300 mg LY) | Part B: C3-C6 (SS/AS + Placebo)
Started | 3 | 2 | 3 | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 3 | 2 | 2 | 2 | 3 | 3 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 2 | 2 | 2 | 3 | 3 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Positive Urine Drug Screen (UDS) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part A Fourth Intervention
Arm/Group | Part A: Cohort 1(C1), Sequence 1 | Part A: C1, Sequence 2 | Part A: C1, Sequence 3 | Part A: Cohort 2 (C2), Sequence 1 | Part A: C2, Sequence 2 | Part A: C2, Sequence 3 | Part B: C3 (Simvastatin [SS]/Atorvastatin[AS] + 5 mg LY) | Part B: C4 (SS/AS + 20 mg LY) | Part B: C5 (SS/AS + 100 mg LY) | Part B: C6 (SS/AS + 300 mg LY) | Part B: C3-C6 (SS/AS + Placebo)
Started | 4 (An additional participant replaced a discontinued participant.) | 2 | 3 (An additional participant replaced a discontinued participant.) | 2 | 3 | 3 | 0 | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 3 | 2 | 3 | 2 | 3 | 2 | 0 | 0 | 0 | 0 | 0
Completed | 3 | 2 | 3 | 2 | 3 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Positive Urinary Drug Screen (UDS) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Part B (Overall)
Arm/Group | Part A: Cohort 1(C1), Sequence 1 | Part A: C1, Sequence 2 | Part A: C1, Sequence 3 | Part A: Cohort 2 (C2), Sequence 1 | Part A: C2, Sequence 2 | Part A: C2, Sequence 3 | Part B: C3 (Simvastatin [SS]/Atorvastatin[AS] + 5 mg LY) | Part B: C4 (SS/AS + 20 mg LY) | Part B: C5 (SS/AS + 100 mg LY) | Part B: C6 (SS/AS + 300 mg LY) | Part B: C3-C6 (SS/AS + Placebo)
Started | 0 (Part A participants completed period 4 and were not in part B.) | 0 (Part A participants completed period 4 and were not in part B.) | 0 (Part A participants completed period 4 and were not in part B.) | 0 (Part A participants completed period 4 and were not in part B.) | 0 (Part A participants completed period 4 and were not in part B.) | 0 (Part A participants completed period 4 and were not in part B.) | 8 (Part B participants randomized to receive 5 mg of LY3202328 + atorvastatin/simvastatin.) | 8 (Part B participants randomized to receive 20 mg of LY3202328 + atorvastatin/simvastatin.) | 8 (Part B participants randomized to receive 100 mg of LY3202328 + atorvastatin/simvastatin.) | 8 (Part B participants randomized to receive 300 mg of LY3202328 + atorvastatin/simvastatin.) | 8 (Part B participants randomized to receive placebo instead of LY3202328 + atorvastatin/simvastatin.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 7 | 8 | 6 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug in Part A and Part B.
Groups:
- Part A, C1, Sequence 1: 1 mg of LY3202328 (LY) was taken orally first intervention, then 10 mg of LY was taken orally second intervention, then placebo was taken orally third intervention, then 600 mg of LY was taken orally fourth intervention.
  C1, Sequence 1:
  (1 mg LY, 10 mg LY, Placebo, 600 mg LY)
- Part A, C1, Sequence 2: 1 mg of LY was taken orally first intervention, then placebo was taken orally second intervention, then 100 mg of LY was taken orally third intervention, then 600 mg of LY was taken orally fourth intervention.
  C1, Sequence 2:
  (1 mg LY, Placebo, 100 mg LY, 600 mg LY)
- Part A, C1, Sequence 3: Placebo was taken orally first intervention, then 10 mg LY was taken orally second intervention, then, 100 mg LY was taken orally third intervention, then placebo was taken orally fourth intervention.
  C1, Sequence 3: (Placebo, 10 mg LY, 100 mg LY, Placebo)
- Part A, C2, Sequence 1: 3 mg of LY was taken orally first intervention, then 30 mg of LY was taken orally second intervention, then placebo was taken orally third intervention, then 30 mg of LY fed was taken orally fourth intervention
  C2, Sequence 1:
  3 mg LY, 30 mg LY, Placebo, 30 mg LY Fed
- Part A, C2, Sequence 2: 3 mg of LY was taken orally first intervention, then placebo was taken orally second intervention, then 300 mg of LY was taken orally third intervention, then placebo was taken orally fourth intervention.
  C2, Sequence 2:
  3 mg LY, Placebo, 300 mg LY, Placebo
- Part A, C2, Sequence 3: Placebo was taken orally first intervention, then 30 mg of LY was taken orally second intervention, then 300 mg of LY was taken orally third intervention, then 30 mg of LY fed was taken orally fourth intervention.
  C2, Sequence 3:
  Placebo, 30 mg LY, 300 mg LY, 30 mg LY Fed
- Part B: SS/AS/Placebo: Participants were randomly assigned to multiple ascending doses of placebo instead of LY at up to 4 dose levels, orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29.
- Part B: SS/AS/5 mg LY: 5 mg of LY was taken orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29.
- Part B: SS/AS/20 mg LY: 20 mg of LY was taken orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29.
- Part B: SS/AS/100 mg LY: 100 mg of LY was taken orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29.
- Part B: SS/AS/300 mg LY: 300 mg of LY was taken orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29.
- Total: Total of all reporting groups
Arm/Group | Part A, C1, Sequence 1 | Part A, C1, Sequence 2 | Part A, C1, Sequence 3 | Part A, C2, Sequence 1 | Part A, C2, Sequence 2 | Part A, C2, Sequence 3 | Part B: SS/AS/Placebo | Part B: SS/AS/5 mg LY | Part B: SS/AS/20 mg LY | Part B: SS/AS/100 mg LY | Part B: SS/AS/300 mg LY | Total
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 3 | 3 | 8 | 8 | 8 | 8 | 8 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.3 (8.02) | 56.0 (12.12) | 58.5 (4.04) | 34.0 (13.53) | 38.3 (22.50) | 54.7 (17.21) | 54.0 (9.12) | 50.5 (12.76) | 46.8 (13.13) | 55.0 (10.18) | 36.9 (10.80) | 48.7 (13.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 0 | 0 | 1 | 4 | 4 | 3 | 4 | 1 | 21
  Male | 3 | 2 | 2 | 3 | 3 | 2 | 4 | 4 | 5 | 4 | 7 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 0 | 0 | 7 | 2 | 15
  Not Hispanic or Latino | 4 | 3 | 4 | 2 | 3 | 3 | 3 | 8 | 8 | 1 | 6 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 3 | 2 | 1 | 1 | 2 | 0 | 0 | 0 | 13
  White | 2 | 2 | 3 | 0 | 1 | 2 | 7 | 6 | 8 | 8 | 8 | 47
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 3 | 4 | 3 | 3 | 3 | 8 | 8 | 8 | 8 | 8 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration Part A and Part B
Description: Number of participants with one or more SAEs in Part A and Part B. A summary of other non-serious adverse events and all serious adverse events, regardless of causality, is located in the Reported Adverse Events Section.
Time Frame: Baseline, Up to 42 Days
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: participants
Groups:
- Part A: Placebo: Participants were randomly assigned to placebo instead of LY in one of the first three periods.
- Part A: 1 mg LY3202328 (LY): 1 mg of LY was taken orally in one of four periods.
- Part A: 3 mg LY: 3 mg of LY was taken orally in one of four periods.
- Part A: 10 mg LY: 10 mg of LY was taken orally in one of four periods.
- Part A: 30 mg LY: 30 mg of LY was taken orally in one of four periods.
- Part A: 100 mg LY: 100 mg of LY was taken orally in one of four periods.
- Part A: 300 mg LY: 300 mg of LY was taken orally in one of four periods.
- Part A: 30 mg LY Fed: 30 mg (fed) of LY was taken orally in one of four periods.
- Part A: 600 mg LY: 600 mg of LY was taken orally in one of four periods.
- Part B: SS/AS/5 mg of LY: 5 mg of LY was taken orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29.
- Part B: SS/AS/20 mg of LY: 20 mg of LY was taken orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29.
- Part B: SS/AS/100 mg of LY: 100 mg of LY was taken orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29.
- Part B: SS/AS/300 mg of LY: 300 mg of LY was taken orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29.
Arm/Group | Part A: Placebo | Part A: 1 mg LY3202328 (LY) | Part A: 3 mg LY | Part A: 10 mg LY | Part A: 30 mg LY | Part A: 100 mg LY | Part A: 300 mg LY | Part A: 30 mg LY Fed | Part A: 600 mg LY | Part B: SS/AS/Placebo | Part B: SS/AS/5 mg of LY | Part B: SS/AS/20 mg of LY | Part B: SS/AS/100 mg of LY | Part B: SS/AS/300 mg of LY
Number analyzed (Participants) | 20 | 7 | 6 | 8 | 6 | 7 | 6 | 7 | 7 | 8 | 8 | 8 | 8 | 8
participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Plasma Concentration (Cmax) of LY3202328 (LY) in Part A After a Single Dose
Description: Pharmacokinetics (PK) is the maximum plasma concentration (Cmax) of LY3202328 Part A after a single dose.
Time Frame: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96 hours Postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data in Part A after a single dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Groups:
- Part A: 1 mg LY: 1 mg of LY was taken orally in one of four periods.
- Part A: 30 mg LY Fed: 30 mg of LY (fed) was taken orally in one of four periods.
Arm/Group | Part A: 1 mg LY | Part A: 3 mg LY | Part A: 10 mg LY | Part A: 30 mg LY | Part A: 100 mg LY | Part A: 300 mg LY | Part A: 600 mg LY | Part A: 30 mg LY Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 4 | 6 | 5 | 4
nanogram/milliliter (ng/mL) | 48.258 (21.11) | 105.023 (26.66) | 340.829 (28.99) | 581.782 (32.29) | 1600.953 (40.01) | 1632.595 (42.84) | 2866.855 (51.29) | 1105.999 (18.47)
Statistical Analysis 1: Comparison: Part A: 30 mg LY vs Part A: 30 mg LY Fed; Geometric Mean Fed/Fasted Ratio of LY3202328 Cmax at 30 mg; Test type: Non-Inferiority — Analyses were based on a pre-defined non-inferiority margin; Least Square Means Percentage = 204.8, 90% CI 2-sided [161.9 to 259.0] — Analysis was the estimate of the ratio fasted versus fed

3. Secondary Outcome: PK: Steady State Maximum Plasma Concentration (Cmax) of LY3202328 (LY) in Part B
Description: PK is the maximum plasma concentration of LY3202328 (Cmax) at steady state in Part B.
Time Frame: Day 28: Predose, 0.5, 1, 2, 4, 4.5, 5, 6, 8, 12, 24 hours Postdose
Population: All randomized participants who received at least one dose of study drug in Part B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Groups:
- Part B: 5 mg LY: 5 mg of LY taken orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29.
- Part B: 20 mg LY: 20 mg of LY taken orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29.
- Part B: 100 mg LY: 100 mg of LY taken orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29.
- Part B: 300 mg LY: 300 mg of LY taken orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29.
Arm/Group | Part B: 5 mg LY | Part B: 20 mg LY | Part B: 100 mg LY | Part B: 300 mg LY
Number analyzed (Participants) | 7 | 8 | 8 | 8
ng/ml | 445.858 (32.78) | 882.125 (32.81) | 3687.167 (34.83) | 3209.396 (37.31)

4. Secondary Outcome: PK: Area Under the Serum Concentration Time Curve From Zero to Infinity (AUC[0-∞]) of LY3202328 (LY) in Part A After a Single Dose
Description: PK is the area under the serum concentration time curve from zero to Infinity (AUC[0-∞]) of LY3202328 in Part A after a single dose.
Time Frame: Day 1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96 hours Postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part A: 3 mg of LY: 3 mg of LY was taken orally in one of four periods.
- Part A: 100 mg of LY: 100 mg of LY was taken orally in one of four periods.
- Part A: 30 mg LY Fed: 30 mg of LY was taken orally in one of four periods.
Arm/Group | Part A: 1 mg LY | Part A: 3 mg of LY | Part A: 10 mg LY | Part A: 30 mg LY | Part A: 100 mg of LY | Part A: 300 mg LY | Part A: 600 mg LY | Part A: 30 mg LY Fed
Number analyzed (Participants) | 1 | 3 | 6 | 6 | 4 | 6 | 2 | 4
ng/mL | NA (NA) — Geometric mean/Coefficient Variation (CV) was not calculated due to n=1. Minimum and maximum values = 1607.0, 1607.0. | NA (NA) — Geometric mean/CV was not calculated due to small sample size n=3. Minimum and maximum values = 2632.0, 3047.0 | 7726.17 (45.23) | 17018.43 (62.60) | 55406.24 (41.35) | 66185.70 (71.44) | NA (NA) — Geometric mean/CV was not calculated due to n=2. Minimum and maximum values = 63062.0, 83978.0. | 28415.22 (56.67)
Statistical Analysis 1: Comparison: Part A: 30 mg LY vs Part A: 30 mg LY Fed; Geometric Mean Fed/Fasted Ratio of LY3202328 AUC(0-inf) at 30 mg; Test type: Non-Inferiority — Analyses were based on a pre-defined non-inferiority margin; Least Squares Mean Percentage = 193.3, 90% CI 2-sided [144.7 to 258.2]

5. Secondary Outcome: PK: Steady State Area Under the Serum Concentration-Time Curve During the Dosing Interval (AUCτ) of LY3202328 (LY) in Part B
Description: PK is the area under the serum concentration-time curve (AUCτ) of LY3202328 at steady state during the dosing interval in Part B.
Time Frame: Day 28: Predose, 0.5, 1, 2, 4, 4.5, 5, 6, 8, 12, 24 hours Postdose
Population: All randomized participants who received at least one dose of study drug in Part B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/milliliter(hr*ng/ml)
Arm/Group | Part B: 5 mg LY | Part B: 20 mg LY | Part B: 100 mg LY | Part B: 300 mg LY
Number analyzed (Participants) | 7 | 8 | 8 | 8
hour*nanogram/milliliter(hr*ng/ml) | 7587.24 (38.612) | 13362.44 (44.984) | 67499.80 (37.465) | 50774.85 (43.861)

6. Secondary Outcome: PK: Time to Maximum Concentration (Tmax) of LY3202328 (LY) in Part A
Description: PK is the time to maximum concentration (Tmax) of LY3202328 in Part A
Time Frame: Day 1: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96 hours Postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data in Part A.
Measure: Median (Full Range); unit: hour (hr)
Groups:
- Part A: 10 mg LY: 10 mg of LY or placebo was taken orally in one of four periods.
Arm/Group | Part A: 1 mg LY | Part A: 3 mg LY | Part A: 10 mg LY | Part A: 30 mg LY | Part A: 100 mg LY | Part A: 300 mg LY | Part A: 600 mg LY | Part A: 30 mg LY Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 4 | 6 | 5 | 4
hour (hr) | 2.02 [1.0 to 4.0] | 3.52 [2.0 to 6.2] | 4.0 [2.0 to 6.0] | 4.00 [3.0 to 4.1] | 6.00 [2.0 to 8.0] | 4.02 [3.0 to 8.0] | 4.00 [2.0 to 24.0] | 5.00 [4.0 to 8.0]

7. Secondary Outcome: PK: Steady State Tmax of LY3202328 (LY) in Part B
Description: PK is the Tmax of LY3202328 at steady state in Part B.
Time Frame: Day 28: Predose, 0.5, 1, 2, 4, 4.5, 5, 6, 8, 12, 24 hours Postdose
Population: All randomized participants who received at least one dose of study drug in Part B.
Measure: Median (Full Range); unit: hr
Arm/Group | Part B: 5 mg LY | Part B: 20 mg LY | Part B: 100 mg LY | Part B: 300 mg LY
Number analyzed (Participants) | 7 | 8 | 8 | 8
hr | 2.00 [2.0 to 6.0] | 4.20 [4.0 to 6.0] | 3.00 [2.0 to 4.0] | 3.04 [1.0 to 6.0]

8. Secondary Outcome: Pharmacodynamics (PD): Change From Baseline in Fasting High-Density Lipoprotein Cholesterol (HDL-c) in Part A
Description: Pharmacodynamics (PD) is the change from Baseline in Fasting High-Density Lipoprotein Cholesterol (HDL-c) in Part A.
Time Frame: Predose, 24, 48, 96 Hours Postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable fasting HDL-c data in Part A.
Measure: Mean (Standard Deviation); unit: millimole/Liter (mmol/L)
Arm/Group | Part A: Placebo | Part A: 1 mg LY | Part A: 3 mg LY | Part A: 10 mg LY | Part A: 30 mg LY | Part A: 100 mg LY | Part A: 300 mg LY | Part A: 600 mg LY
Number analyzed (Participants) | 19 | 6 | 6 | 5 | 6 | 6 | 5 | 5
millimole/Liter (mmol/L)
  24 Hours | -0.003 (0.1155) | -0.030 (0.0842) | -0.043 (0.0454) | -0.047 (0.0740) | -0.026 (0.0433) | 0.052 (0.1099) | -0.004 (0.0684) | 0.010 (0.0232)
  48 Hours | -0.037 (0.1560) | -0.039 (0.0217) | 0.009 (0.1387) | -0.043 (0.0950) | -0.026 (0.1010) | 0.019 (0.0978) | -0.009 (0.1551) | -0.052 (0.0755)
  96 Hours | -0.074 (0.1258) | -0.073 (0.1241) | -0.086 (0.0892) | -0.134 (0.0553) | -0.030 (0.1304) | -0.091 (0.1206) | -0.082 (0.1487) | -0.005 (0.1411)

9. Secondary Outcome: PD: Change From Baseline to Last Day of Dosing in Fasting HDL-c in Part B
Description: PD is the change from baseline to last day of dosing in fasting HDL-c in Part B.
Time Frame: Predose, Days 7, 14, 21, and 28 Postdose
Population: All randomized participants who received at least one dose of study drug in Part B.
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Part B: Placebo: A multiple ascending dose of placebo instead of LY at up to 4 dose levels, orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29.
- Part B: 300 mg LY: 300 mg of LY taken orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) week prior to treatment and on Day 29.
Arm/Group | Part B: Placebo | Part B: 5 mg LY | Part B: 20 mg LY | Part B: 100 mg LY | Part B: 300 mg LY
Number analyzed (Participants) | 8 | 7 | 8 | 8 | 8
mmol/L | 0.008 (0.1169) | -0.010 (0.1165) | -0.101 (0.0812) | -0.107 (0.1894) | -0.101 (0.0621)

10. Secondary Outcome: PD: Change From Baseline in Fasting Total Triglycerides Part A
Description: PD is the change from baseline in fasting total triglycerides in Part A.
Time Frame: Predose, 24, 48, 96 Hours Postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable fasting triglyceride data in Part A.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part A: Placebo | Part A: 1 mg LY | Part A: 3 mg LY | Part A: 10 mg LY | Part A: 30 mg LY | Part A: 100 mg LY | Part A: 300 mg LY | Part A: 600 mg LY
Number analyzed (Participants) | 19 | 6 | 6 | 5 | 6 | 6 | 5 | 5
mmol/L
  24 Hours | -0.276 (0.2043) | -0.397 (0.2877) | -0.190 (0.1491) | -0.386 (0.2766) | -0.311 (0.2831) | -0.523 (0.5801) | -0.064 (0.1455) | -0.302 (0.2318)
  48 Hours | -0.320 (0.3162) | -0.269 (0.2260) | -0.115 (0.2643) | -0.260 (0.3382) | -0.418 (0.3290) | -0.766 (0.5870) | -0.226 (0.3646) | -0.198 (0.1345)
  96 Hours | -0.239 (0.3227) | -0.209 (0.6817) | -0.132 (0.2349) | 0.013 (0.7179) | -0.331 (0.4343) | -0.455 (0.5144) | -0.326 (0.3549) | 0.158 (0.6773)

11. Secondary Outcome: PD: Change From Baseline to Last Day of Dosing in Fasting Total Triglycerides in Part B
Description: PD is the change from baseline to last day of dosing in fasting total triglycerides in Part B.
Time Frame: Predose, Days 7, 14, 21, and 28 Postdose
Population: All randomized participants who received at least one dose of study drug in Part B.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part B: Placebo | Part B: 5 mg LY | Part B: 20 mg LY | Part B: 100 mg LY | Part B: 300 mg LY
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
mmol/L | 0.205 (0.6757) | -0.131 (0.2720) | -0.231 (0.5383) | 0.020 (0.6281) | -0.480 (0.5235)

12. Secondary Outcome: PD: Change From Baseline to in Fasting Total Cholesterol in Part A
Description: PD is the change from baseline in fasting total cholesterol in Part A.
Time Frame: Predose, 24, 28, 96 Hours Postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable fasting total cholesterol data in Part A.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part A: Placebo | Part A: 1 mg LY | Part A: 3 mg LY | Part A: 10 mg LY | Part A: 30 mg LY | Part A: 100 mg LY | Part A: 300 mg LY | Part A: 600 mg LY
Number analyzed (Participants) | 19 | 6 | 6 | 5 | 6 | 4 | 6 | 5
mmol/L
  24 Hours | 0.085 (0.3075) | -0.186 (0.2699) | -0.013 (0.2850) | -0.203 (0.2157) | 0.073 (0.1863) | 0.285 (0.1903) | 0.203 (0.2421) | 0.093 (0.1560)
  48 Hours | -0.085 (0.4618) | -0.436 (0.2608) | -0.030 (0.2218) | -0.376 (0.2321) | -0.013 (0.3981) | 0.091 (0.3654) | 0.134 (0.5446) | -0.026 (0.4719)
  96 Hours | -0.318 (0.4288) | -0.527 (0.3262) | -0.207 (0.2949) | -0.609 (0.2635) | -0.199 (0.4732) | -0.317 (0.6296) | -0.155 (0.4826) | -0.041 (0.6020)

13. Secondary Outcome: PD: Change From Baseline to Last Day of Dosing in Fasting Total Cholesterol in Part B
Description: PD is the change from baseline to last day of dosing in fasting total cholesterol in Part B.
Time Frame: Predose, Days 7, 14, 21, and 28 Postdose
Population: All randomized participants who received at least one dose of study drug in Part B.
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Part B: Placebo: A multiple ascending dose of placebo at up to 4 dose levels, orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29.
Arm/Group | Part B: Placebo | Part B: 5 mg LY | Part B: 20 mg LY | Part B: 100 mg LY | Part B: 300 mg LY
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
mmol/L | 0.206 (0.3615) | 0.118 (0.3840) | 0.183 (0.4681) | 0.174 (0.4963) | -0.190 (0.4425)

14. Secondary Outcome: PD: Change From Baseline in Fasting Low-Density Lipoprotein Cholesterol (LDL-c) in Part A
Description: PD is the change from baseline in fasting low-density lipoprotein cholesterol (LDL-c) Part A.
Time Frame: Predose, 24, 48, 96 Hours Postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable LDL-c data in Part A.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Part A: Placebo | Part A: 1 mg LY | Part A: 3 mg LY | Part A: 10 mg LY | Part A: 30 mg LY | Part A: 100 mg LY | Part A: 300 mg LY | Part A: 600 mg LY
Number analyzed (Participants) | 19 | 6 | 6 | 5 | 6 | 6 | 5 | 5
mmol/L
  24 Hours | 0.231 (0.2513) | 0.025 (0.2205) | 0.117 (0.2400) | 0.020 (0.2328) | 0.241 (0.1594) | 0.471 (0.3418) | 0.236 (0.2429) | 0.163 (0.1608)
  48 Hours | 0.111 (0.4026) | -0.275 (0.3004) | 0.013 (0.2093) | -0.214 (0.2378) | 0.203 (0.3400) | 0.419 (0.3293) | 0.245 (0.3457) | -0.001 (0.3891)
  96 Hours | -0.109 (0.4147) | -0.358 (0.4170) | -0.061 (0.1747) | -0.481 (0.3681) | -0.018 (0.3048) | -0.020 (0.6327) | 0.075 (0.2565) | 0.038 (0.6305)

15. Secondary Outcome: PD: Change From Baseline to Last Day of Dosing in Fasting LDL-c in Part B
Description: PD is the change from baseline to last day of dosing in fasting LDL-c in Part B.
Time Frame: Predose, Days 7, 14, 21, and 28 Postdose
Population: All randomized participants who received at least one dose of study in Part B.
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Part B: Placebo: Participants were randomly assigned to multiple ascending doses of placebo instead of LY at up to 4 dose levels, orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29.
- Part B: 300 mg LY: 5 mg of LY taken orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29.
Arm/Group | Part B: Placebo | Part B: 5 mg LY | Part B: 20 mg LY | Part B: 100 mg LY | Part B: 300 mg LY
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
mmol/L | 0.103 (0.4114) | 0.184 (0.3419) | 0.388 (0.4876) | 0.227 (0.4494) | 0.131 (0.4225)

16. Secondary Outcome: PK: Cmax of Simvastatin With/Without LY3202328 (LY) in Part B
Description: PK: Cmax of Simvastatin with/without LY3202328 (LY) Co-administration in Part B.
Time Frame: Day -7 and Day 28: Predose, 0.5, 1, 2, 4, 4.5, 5, 6, 8, 12, 24 hours Postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data in Part B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Groups:
- Simvastatin With LY (Test): A single simvastatin test dose was taken fasted a week prior to LY treatment initiation, and on Day 29 after initiation of LY daily dosing (coadministered with LY).
- Simvastatin Alone (Reference): A single simvastatin reference dose was taken fasted a week prior to LY treatment initiation, and on Day 29 after initiation of LY daily dosing without LY.
Arm/Group | Simvastatin With LY (Test) | Simvastatin Alone (Reference)
Number analyzed (Participants) | 8 | 8
ng/ml
  Placebo | 2.906 (18.72) | 2.061 (71.24)
  5 mg LY | 2.388 (58.17) | 3.374 (52.99)
  20 mg LY | 3.576 (19.35) | 3.274 (26.87)
  100 mg LY | 4.634 (55.59) | 4.303 (25.45)
  300 mg LY | 4.221 (58.78) | 1.979 (55.84)
Statistical Analysis 1: Comparison: Simvastatin With LY (Test) vs Simvastatin Alone (Reference); Part B Placebo; Test type: Other — Ratio estimate without hypothesis testing; Geometric Least Square Means Ratio (%) = 141.0, 90% CI 2-sided [67.9 to 293.0]
Statistical Analysis 2: Comparison: Simvastatin With LY (Test) vs Simvastatin Alone (Reference); Part B 5 mg LY; Test type: Other — Ratio estimate without hypothesis testing; Geometric Least Square Means Ratio (%) = 70.8, 90% CI 2-sided [31.9 to 157.1]
Statistical Analysis 3: Comparison: Simvastatin With LY (Test) vs Simvastatin Alone (Reference); Part B 20 mg LY; Test type: Other — Ratio estimate without hypothesis testing; Geometric Least Square Means Ratio (%) = 109.2, 90% CI 2-sided [99.8 to 119.5]
Statistical Analysis 4: Comparison: Simvastatin With LY (Test) vs Simvastatin Alone (Reference); Part B 100 mg LY; Test type: Other — Ratio estimate without hypothesis testing; Geometric Least Square Means Ratio (%) = 107.7, 90% CI 2-sided [68.1 to 170.4]
Statistical Analysis 5: Comparison: Simvastatin With LY (Test) vs Simvastatin Alone (Reference); Part B 300 mg LY; Test type: Other — Ratio estimate without hypothesis testing; Geometric Least Squares Mean Ratio (%) = 213.3, 90% CI 2-sided [200.3 to 227.1]
Statistical Analysis 6: Comparison: Simvastatin With LY (Test) vs Simvastatin Alone (Reference); Part B Overall; Test type: Other — Ratio estimate without hypothesis testing; Geometric Least Square Means Ratio (%) = 115.4, 90% CI 2-sided [91.2 to 146.2]

17. Secondary Outcome: PK: Area Under Concentration Curve From Zero to Time (AUC [0-t]) of Simvastatin With/Without LY3202328 (LY) in Part B
Description: PK: Area Under Concentration Curve From Zero to Time (AUC [0-t]) of Simvastatin with/without LY3202328 (LY) Co-administration in Part B. AUC from time 0 to time t, where t is the time of last quantifiable plasma concentration.
Time Frame: Day -7 and Day 28: Predose, 0.5, 1, 2, 4, 4.5, 5, 6, 8, 12, 24 hours Postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data in Part B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/ml
Arm/Group | Simvastatin With LY (Test) | Simvastatin Alone (Reference)
Number analyzed (Participants) | 8 | 8
hr*ng/ml
  Placebo | 9.648 (38.82) | 6.250 (61.54)
  5 mg LY | 6.668 (42.96) | 9.287 (57.54)
  20 mg LY | 9.697 (26.81) | 7.960 (32.21)
  100 mg LY | 14.269 (53.78) | 10.434 (26.20)
  300 mg LY | 11.908 (60.19) | 8.951 (61.65)
Statistical Analysis 1: Comparison: Simvastatin With LY (Test) vs Simvastatin Alone (Reference); Part B Placebo; Test type: Other — Ratio estimate without hypothesis testing; Geometric Least Squares Mean Ratio (%) = 155, 90% CI 2-sided [87.6 to 274.2]
Statistical Analysis 2: Comparison: Simvastatin With LY (Test) vs Simvastatin Alone (Reference); Part B 5 mg LY; Test type: Other — Ratio estimate without hypothesis testing; Geometric Least Squares Mean Ratio (%) = 71.5, 90% CI 2-sided [40.7 to 125.3]
Statistical Analysis 3: Comparison: Simvastatin With LY (Test) vs Simvastatin Alone (Reference); Part B 20 mg LY; Test type: Other — Ratio estimate without hypothesis testing; Geometric Least Squares Mean Ratios (%) = 122.4, 90% CI 2-sided [90.7 to 165.1]
Statistical Analysis 4: Comparison: Simvastatin With LY (Test) vs Simvastatin Alone (Reference); Part B 100 mg LY; Test type: Other — Ratio estimate without hypothesis testing; Geometric Least Squares Mean Ratio (%) = 136.6, 90% CI 2-sided [89.8 to 207.7]
Statistical Analysis 5: Comparison: Simvastatin With LY (Test) vs Simvastatin Alone (Reference); Part B 300 mg LY; Test type: Other — Ratio estimate without hypothesis testing; Geometric Least Squares Mean Ratio (%) = 132.6, 90% CI 2-sided [90.5 to 194.4]
Statistical Analysis 6: Comparison: Simvastatin With LY (Test) vs Simvastatin Alone (Reference); Part B Overall; Test type: Other — Ratio estimate without hypothesis; Geometric Least Squares Mean Ratio (%) = 112.2, 90% CI 2-sided [93.2 to 135.1]

18. Secondary Outcome: PK: Cmax of Atorvastatin With/Without LY3202328 (LY) in Part B
Description: PK: Cmax of Atorvastatin with/without LY3202328 (LY) Co-administration in Part B.
Time Frame: Day -7 and Day 28: Predose, 0.5, 1, 2, 4, 4.5, 5, 6, 8, 12, 24 hours Postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data in Part B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Atorvastatin With LY (Test): A single atorvastatin test dose was taken fasted a week prior to LY treatment initiation, and on Day 29 after initiation of LY daily dosing (coadministered with LY).
- Atorvastatin Alone (Reference): A single atorvastatin reference dose was taken fasted a week prior to LY treatment initiation, and on Day 29 after initiation of LY daily dosing without LY.
Arm/Group | Atorvastatin With LY (Test) | Atorvastatin Alone (Reference)
Number analyzed (Participants) | 8 | 8
ng/mL
  Placebo | 3.479 (20.58) | 3.575 (30.44)
  5 mg LY | 2.840 (27.96) | 3.621 (82.05)
  20 mg LY | 1.238 (38.05) | 1.286 (45.27)
  100 mg LY | 2.511 (32.17) | 3.105 (51.95)
  300 mg LY | 1.489 (42.11) | 1.376 (59.68)
Statistical Analysis 1: Comparison: Atorvastatin With LY (Test) vs Atorvastatin Alone (Reference); Part B Placebo; Test type: Other — Ratio estimate without hypothesis testing; Geometric Least Squares Mean Ratio (%) = 97.3, 90% CI 2-sided [80.4 to 117.8]
Statistical Analysis 2: Comparison: Atorvastatin With LY (Test) vs Atorvastatin Alone (Reference); Test type: Other — Ratio estimate without hypothesis testing; Geometric Least Squares Mean Ratio (%) = 57.5, 90% CI 2-sided [31.3 to 106.0]
Statistical Analysis 3: Comparison: Atorvastatin With LY (Test) vs Atorvastatin Alone (Reference); Part B 20 mg LY; Test type: Other — Ratio estimate without hypothesis testing; Geometric Least Squares Mean Ratio (%) = 96.2, 90% CI 2-sided [66.8 to 138.7]
Statistical Analysis 4: Comparison: Atorvastatin With LY (Test) vs Atorvastatin Alone (Reference); Part B 100 mg LY; Test type: Other — Ratio estimate without hypothesis testing; Geometric Least Squares Mean Ratio (%) = 80.9, 90% CI 2-sided [45.8 to 142.7]
Statistical Analysis 5: Comparison: Atorvastatin With LY (Test) vs Atorvastatin Alone (Reference); Part B 300 mg LY; Test type: Other — Ratio estimate without hypothesis testing; Geometric Least Squares Mean Ratio (%) = 108.2, 90% CI 2-sided [40.2 to 291.2]
Statistical Analysis 6: Comparison: Atorvastatin With LY (Test) vs Atorvastatin Alone (Reference); Part B Overall; Test type: Other — Ratio estimate without hypothesis; Geometric Least Squares Mean Ratio (%) = 87.9, 90% CI 2-sided [67.4 to 114.7]

19. Secondary Outcome: PK: AUC (0-t) of Atorvastatin With/Without LY3202328 (LY) in Part B
Description: PK: AUC (0-t) of Atorvastatin with/without LY3202328 (LY) Co-administration in Part B. AUC from time 0 to time t, where t is the time of last quantifiable plasma concentration.
Time Frame: Day -7 and Day 28: Predose, 0.5, 1, 2, 4, 4.5, 5, 6, 8, 12, 24 hours Postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data in Part B.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/ml
Arm/Group | Atorvastatin With LY (Test) | Atorvastatin Alone (Reference)
Number analyzed (Participants) | 8 | 8
hr*ng/ml
  Placebo | 15.874 (32.81) | 16.518 (33.88)
  5 mg LY | 17.311 (6.35) | 14.913 (48.97)
  20 mg LY | 7.921 (57.94) | 7.952 (63.04)
  100 mg LY | 11.983 (38.63) | 13.207 (61.25)
  300 mg LY | 7.748 (50.04) | 9.111 (36.39)
Statistical Analysis 1: Comparison: Atorvastatin With LY (Test) vs Atorvastatin Alone (Reference); Part B Placebo; Test type: Other — Ratio estimate without hypothesis testing; Geometric Least Square Means Ratio (%) = 96.0, 90% CI 2-sided [90.2 to 102.1]
Statistical Analysis 2: Comparison: Atorvastatin With LY (Test) vs Atorvastatin Alone (Reference); Part B 5 mg LY; Test type: Other — Ratio estimate without hypothesis testing; Geometric Least Squares Mean Ratio (%) = 90.7, 90% CI 2-sided [59.8 to 137.6]
Statistical Analysis 3: Comparison: Atorvastatin With LY (Test) vs Atorvastatin Alone (Reference); Part B 20 mg LY; Test type: Other — Ratio estimate without hypothesis testing; Geometric Least Square Means Ratio (%) = 99.9, 90% CI 2-sided [75.9 to 131.5]
Statistical Analysis 4: Comparison: Atorvastatin With LY (Test) vs Atorvastatin Alone (Reference); Part B 100 mg LY; Test type: Other — Ratio estimate without hypothesis testing; Geometric Least Square Means Ratio (%) = 91.0, 90% CI 2-sided [67.5 to 122.7]
Statistical Analysis 5: Comparison: Atorvastatin With LY (Test) vs Atorvastatin Alone (Reference); Part B 300 mg LY; Test type: Other — Ratio estimate without hypothesis testing; Geometric Least Squares Mean Ratio (%) = 87.0, 90% CI 2-sided [42.0 to 180.5]
Statistical Analysis 6: Comparison: Atorvastatin With LY (Test) vs Atorvastatin Alone (Reference); Part B Overall; Test type: Other — Ratio estimate without hypothesis; Geometric Least Squares Mean Ratio (%) = 93.5, 90% CI 2-sided [81.8 to 106.9]

ADVERSE EVENTS:
Time Frame: From Baseline to End of Study (Up to 10 Weeks)
Description: The safety population are all participants part A and part B combined who received at least one dose of study drug. Several participants received placebo for a second time during the fourth dosing interval, so these participants had 2 placebo-dosing periods.
Groups:
- Placebo: Participants were randomly assigned to placebo instead of LY in one of the first three periods in Part A. Participants were randomly assigned to multiple ascending doses of placebo instead of LY at up to 4 dose levels, orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29 in Part B.
- 1 mg LY3202328 (LY): 1 mg of LY was taken orally in one of four periods in Part A.
- 3 mg LY: 3 mg of LY was taken orally in one of four periods in Part A.
- 5 mg LY: 5 mg of LY was taken orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29 in Part B.
- 10 mg LY: 10 mg of LY was taken orally in one of four periods in Part A.
- 20 mg LY: 20 mg of LY was taken orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29 in Part B.
- 30 mg LY: 30 mg of LY was taken orally in one of four periods in Part A.
- 30 mg LY Fed: 30 mg of LY (fed) was taken orally in one of four periods in Part A.
- 100 mg LY: 100 mg of LY was taken orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29 in Part B.
- 300 mg LY: 300 mg of LY was taken orally, once daily for 29 days, while fasting and with a single dose of 10 mg statin (SS/AS) one week prior to treatment and on Day 29 in Part B.
- 600 mg of LY: 600 mg of LY was taken orally in one of four periods in Part A.
Arm/Group | Placebo | 1 mg LY3202328 (LY) | 3 mg LY | 5 mg LY | 10 mg LY | 20 mg LY | 30 mg LY | 30 mg LY Fed | 100 mg LY | 300 mg LY | 600 mg of LY
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/6 | 0/6 | 0/8 | 0/6 | 0/8 | 0/6 | 0/4 | 0/12 | 0/14 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/6 | 0/6 | 0/8 | 0/6 | 0/8 | 0/6 | 0/4 | 0/12 | 2/14 | 0/5
Other Adverse Events (participants affected / at risk) | 2/25 | 0/6 | 0/6 | 5/8 | 2/6 | 5/8 | 1/6 | 0/4 | 1/12 | 6/14 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=25) | 1 mg LY3202328 (LY) (N=6) | 3 mg LY (N=6) | 5 mg LY (N=8) | 10 mg LY (N=6) | 20 mg LY (N=8) | 30 mg LY (N=6) | 30 mg LY Fed (N=4) | 100 mg LY (N=12) | 300 mg LY (N=14) | 600 mg of LY (N=5)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=25) | 1 mg LY3202328 (LY) (N=6) | 3 mg LY (N=6) | 5 mg LY (N=8) | 10 mg LY (N=6) | 20 mg LY (N=8) | 30 mg LY (N=6) | 30 mg LY Fed (N=4) | 100 mg LY (N=12) | 300 mg LY (N=14) | 600 mg of LY (N=5)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Alt increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pr interval prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stiff neck (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatographic urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushed (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (3):
  • Study Protocol: GSEA Protocol (2016-01-28): https://cdn.clinicaltrials.gov/large-docs/69/NCT02714569/Prot_000.pdf
  • Study Protocol: GSEA Protocol (a) (2016-06-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT02714569/Prot_001.pdf
  • Statistical Analysis Plan (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/69/NCT02714569/SAP_002.pdf